CLINICAL TRIAL: NCT00627367
Title: A Randomized Controlled Trial Comparing Protocolized Versus Non-protocolized Treatment of Adult ED Patients With Acute Severe Pain
Brief Title: Protocolized vs Nonprotocolized Treatment of Adult ED Patients With Acute Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, MD, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC 0710359
Record Dates: First submitted 2008-02-21; First posted 2008-03-03 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Acute Pain
Keywords: Acute Pain, Emergency Department, ED, Hydromorphone, Dilaudid Protocolized Nonprotocolized Usual Care
MeSH Terms: conditions — Acute Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocolized (Experimental): 1mg IV hydromorphone followed by an additional 1mg at 15 minutes if the patient answer "yes" to the question, "Do you want more pain medication?"
  Interventions: Drug: Hydromorphone
- Nonprotocolized (Active Comparator): An IV opioid the type and dose of which will be determined by the treating clincian
  Interventions: Drug: Nonprotocolized

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone 1mg IV, followed by an optional dose of 1mg IV hydromorphone 15 minutes
  Other Names: Dilaudid
  Arms: Protocolized
Drug: Nonprotocolized — An IV opioid the type and dose of which will be determined by the treating clinician
  Other Names: Usual Care
  Arms: Nonprotocolized

SUMMARY:
Patients treated with protocolized pain management (1 mg of IV hydromorphone followed by an additional 1 mg IV hydromorphone if the patient wants more) will have better pain relief and no more adverse events than patients receiving non-protocolized pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 64 years: Patients under the age of 21 are automatically triaged to the Children's Hospital at Montefiore Emergency Department, and hence cannot be enrolled in this study. Age 64 was selected as an upper range for inclusion because substantial evidence supports age as being an important determinant of morphine requirement over longer periods of time.
2. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in ED literature.
3. Emergency Department (ED) attending physician's judgment that patient's pain warrants use of intravenous opioids: The factors that influence the decision to use intravenous opioids are complex and extensive. An approach that is commonly taken to address the issue of patient selection in drug trials is to use a specific condition (e.g., renal colic) or treatment (e.g., post-hysterectomy) that would generally be thought to be appropriately treated with an opioid analgesic, thereby eliminating individual judgment about eligibility for the study. However in order to assess the role of intravenous (IV) opioids with the widest generalizability in the ED setting, we decided to enroll patients with a variety of diagnoses, all with a complaint of acute pain. Opioids are not an appropriate treatment for all patients who present with a complaint of pain (e.g., gastroenteritis, migraine). Therefore either a comprehensive list of diagnoses and situations in which opioids are indicated must be specified, or clinical judgment needs to be used. We have opted for the latter alternative.
4. Normal mental status: In order to provide measures of pain experienced the patient needs to have a normal mental status. Orientation to person, place and time will be used as an indicator of sufficiently normal mental status to participate in the study.

Exclusion Criteria:

1. Prior use of methadone: the effect of methadone use on the perception of acute pain is unknown and suspected to be altered.
2. Use of other opioids, tramadol, or heroin in the past seven days: to avoid introducing bias related to opioid tolerance that may alter the response to intravenous opioids thereby masking the effects of the medications administered.
3. Prior adverse reaction to morphine, hydromorphone, or other opioids: An exception will be if the patient has received opioid medications in the past without adverse event (i.e. a patient may state he is allergic to morphine but has received hydromorphone in the past without any adverse effects)
4. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months resulting in alteration in pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, migraine, and peripheral neuropathies.
5. Alcohol intoxication: the presence of alcohol intoxication may alter the perception, report, and treatment of pain. Alcohol intoxication will be determined to exist as judged by the treating physician.
6. Systolic Blood Pressure < 90 mm Hg: Opioids produce peripheral vasodilation that may result in orthostatic hypotension or syncope.
7. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant depression of respiration or coma.
8. Weight less than 100 pounds: we are concerned that hydromorphone in doses up to 2 mg may not be safe in patients weighing less than 100 lbs.
9. Baseline room air oxygen saturation less than 95%: since IV opioids may cause respiratory depression and result in hypoxemia, we are excluding this subgroup of patients.
10. C02 measurement greater than 46: In accordance with a similar study (04-12-360), four subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46, then the patient will be excluded from the study. The 4 subsets are as follows:

    1. All patients who have a history of chronic obstructive pulmonary disease (COPD)
    2. All patients who have a history of sleep apnea
    3. All patients who report a history of asthma together with greater than a 20 pack-year smoking history
    4. All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, M.D., Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protocolized | Nonprotocolized
Started | 112 | 112
Completed | 112 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The difference between the number of participants who enrolled and completed the study and the number of participants analyzed is due to missing outcome data. There were 4 missing data from the Protocolized group, and 2 missing data from the Nonprotocolized group, for a total of 6 patients. These 6 patients were excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocolized | Nonprotocolized | Total
Number analyzed (Participants) | 108 | 110 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11) | 41 (12) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 75 | 141
  Male | 42 | 35 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 25 | 34 | 59
  White | 9 | 8 | 17
  Hispanic | 72 | 66 | 138
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 110 | 218
Weight [Mean (Standard Deviation); unit: lbs] | 179 (52) | 177 (49) | 178 (51)
Location of Pain [Count of Participants; unit: Participants]
  Abdomen | 59 | 73 | 132
  Other | 49 | 37 | 86
Pain Intensity [Count of Participants; unit: Participants] — Pain intensity is measured on a numerical rating score (NRS) scale of 0 ("no pain") to 10 ("worst pain imaginable"). This pain intensity measure is the pain intensity of the patient before treatment in the Emergency Department.
  Participants
    3-7 | 8 | 15 | 23
    8 | 22 | 26 | 48
    9 | 11 | 14 | 25
    10 | 67 | 55 | 122
Nausea/vomiting [Count of Participants; unit: Participants] | 44 | 54 | 98
Analgesics taken at home [Count of Participants; unit: Participants] | 35 | 26 | 61

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Change in Pain Intensity From Initial Administration of Analgesics (Baseline) to 60 Minutes Post-baseline.
Description: Pain intensity is rated on the numerical rating scale (NRS), measured in integer units from 0 ("no pain") to 10 ("worst pain imaginable"). The change in pain intensity subtracts the NRS score given by the patient 60 minutes after treatment was administered from the baseline NRS score (before treatment in the Emergency Department).
Time Frame: 60 minutes
Population: Protocolized group had 4 missing outcome data, Nonprotocolized missing 2 outcome data. These 6 patients were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protocolized | Nonprotocolized
Number analyzed (Participants) | 108 | 110
units on a scale | 5.5 (2.9) | 4.5 (3.0)

2. Post Hoc Outcome: Change in Numerical Rating Scale (NRS) Scores Among Patients Who Received 1 Dose of Intravenous (IV) Hydromorphone
Description: Pain intensity is rated on the numerical rating scale (NRS), measured in integer units from 0 ("no pain") to 10 ("worst pain imaginable"). The change in pain intensity subtracts the NRS score given by the patient 60 minutes after treatment was administered from the baseline score (before treatment in the Emergency Department).
Time Frame: 60 minutes
Population: Change in N from total analyzed (82 and 99 from 108 and 110 respectively) due to looking at a subpopulation: those patients who only received 1 dose of IV hydromorphone, versus those who received 2 or more doses (see 3. Post Hoc Outcome).
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Protocolized | Nonprotocolized
Number analyzed (Participants) | 82 | 99
units on a scale | 6.1 (4.0) | 4.5 (3.1)

3. Post Hoc Outcome: Change in Numerical Rating Scale (NRS) Scores Among Patients Who Received 2 Doses of Intravenous (IV) Hydromorphone
Description: as for outcome 2
Time Frame: 60 minutes
Population: Change in N from total analyzed (26 and 22 from 108 and 110 respectively) due to looking at a subpopulation: those patients who received 2 or more doses of IV hydromorphone, versus those who received only 1 dose (see 2. Post Hoc Outcome).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protocolized | Nonprotocolized
Number analyzed (Participants) | 26 | 11
units on a scale | 4.0 (3.2) | 4.3 (3.3)

4. Post Hoc Outcome: Change in Numerical Rating Scale (NRS) Scores Among Patients in the Protocolized Group vs Those in the Physician Driven Group Who Received Only Intravenous (IV) Morphine
Description: Pain intensity is rated on the numerical rating scale (NRS), measured in integer units from 0 ("no pain") to 10 ("worst pain imaginable"). The change in pain intensity subtracts the NRS score given by the patient 60 minutes after treatment was administered from the baseline score (before treatment in the Emergency Department). The comparison of hydromorphone to morphine is due to the wide use of morphine for pain management in the Emergency Department setting and the comparison of the two opioids in previous studies.
Time Frame: 60 minutes
Population: The Nonprotocolized group has a different value for participants analyzed for this section than the overall number of participants analyzed for the group (81 versus 110), because this is looking at only those patients who received IV morphine. Nonprotocolized left medication up to the doctor, and as such, some patients received different medication
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nonprotocolized: An IV opioid the type and dose of which will be determined by the treating clincian
  Nonprotocolized: An IV opioid the type and dose of which will be determined by the treating clinician. For this subanalysis, only patients who received IV morphine are analyzed
Arm/Group | Protocolized | Nonprotocolized
Number analyzed (Participants) | 108 | 81
units on a scale | 5.6 (3.2) | 4.4 (2.8)

ADVERSE EVENTS:
Time Frame: 60 minutes after the last dose of opioids was given
Arm/Group | Protocolized | Nonprotocolized
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/110
Other Adverse Events (participants affected / at risk) | 33/108 | 27/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Protocolized (N=108) | Nonprotocolized (N=110)
Oxygen saturation <90% (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oxygen saturation 90-94% (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulse rate <60 beats/min (Vascular disorders) | 4/106 | 9/106 — excludes patients with baseline pulse below 60 beats/min
Systolic blood pressure <90 mmHg (Vascular disorders) | 2 | 3/108
Respiratory rate <12 breaths /min (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 11/64 | 5/56 — excludes patients who were nauseated or had vomited before first dose of IV opioid
Vomiting (Gastrointestinal disorders) | 3/64 | 1/56 — excludes patients who were nauseated or had vomited before first dose of IV opioid
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes